CLINICAL TRIAL: NCT01506128
Title: Exploration of Optimal Experimental Settings to Detect Human Papillomavirus From Menstrual Blood in Women With High-grade Squamous Intraepithelial Lesion or High-risk Human Papillomavirus Infection
Brief Title: Human Papillomavirus in Menstrual Blood
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kidong Kim, Assistant Professor, Department of Obstetrics and Gynecology, Seoul National University Bundang Hospital
Other Study IDs: SNUBH_GO_001
Record Dates: First submitted 2012-01-03; First posted 2012-01-09 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Human Papillomavirus
Keywords: HPV; Menstrual blood; HPV detection using menstrual blood

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Menstrual blood in pad
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HPV: Premenopausal women with HSIL in Pap test or high-risk HPV
  Interventions: Other: Collecting a Pad used at the first menstrual period after enrollment

INTERVENTIONS:
Other: Collecting a Pad used at the first menstrual period after enrollment — Collecting a Pad used at the first menstrual period after enrollment

SUMMARY:
The investigators tried to know whether a virus causing cervical cancer could be detected in menstrual blood and to set up a experimental setting to detect the virus.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women with HSIL at Pap test or high-risk HPV

Exclusion Criteria:

* Suspicious cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Premenopausal women with HSIL at Pap test or high-risk HPV
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
HPV detection rate in menstrual blood | First period after enrollment usually within 2 months after enrollment
  The first menstrual period after enrollment is assumed to occur within 2 months. At that time, the participant used pads and send the used pads to investigators. The investigator do procedures to detect HPV in pads.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea